CLINICAL TRIAL: NCT01118286
Title: AdADOSE - Antihypertensive Treatment With Adalat® in Different Doses and Combination Therapy
Brief Title: Treatment of Hypertension With Adalat® in Combination With Other Drugs
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Medical Affairs Therapeutic Area Head, Bayer Healthcare AG
Other Study IDs: 14296; AL0701 (Other: company internal); AdADOSE (Other: company internal)
Record Dates: First submitted 2010-05-05; First posted 2010-05-06 (Estimated); Last update posted 2012-06-27 (Estimated); Status verified 2012-06

CONDITIONS: Hypertension
Keywords: Hypertension; Drug therapy, combination
MeSH Terms: conditions — Hypertension | interventions — Nifedipine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Nifedipine (Adalat, BAYA1040)

INTERVENTIONS:
Drug: Nifedipine (Adalat, BAYA1040) — Previously untreated hypertensive adult patients starting with combination therapy containing nifedipine or insufficiently controlled hypertensive patients receiving nifedipine as an add-on to existing non-CCB containing antihypertensive therapy. The decision of including the patient as well as decision on dosage and duration is taken by the investigator.

SUMMARY:
To investigate the therapeutic effectiveness of long acting nifedipine containing combination therapy in the treatment of hypertensive patients.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated hypertensive patients starting with combination therapy containing nifedipine or
* Insufficiently controlled hypertensive pts. receiving nifedipine as an add-on to existing non-CCB (calcium-channel-blocker) containing antihypertensive therapy

Exclusion Criteria:

* None. Exclusion criteria are defined by contraindications and precautions as stated in the local product information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Previously untreated hypertensive adult patients starting with combination therapy containing nifedipine or insufficiently controlled hypertensive patients receiving nifedipine as an add-on to existing non-CCB containing antihypertensive therapy
Sampling Method: Non-Probability Sample
Enrollment: 4497 (Actual)
Dates: Start 2010-01; Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of treatment success (lowering of blood pressure in mmHg) in adult hypertensive patients | After three months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (11):
- Many Locations, Bahrain
- Many Locations, Egypt
- Many Locations, Jordan
- Many Locations, Lebanon
- Many Locations, Morocco
- Many Locations, Oman
- Many Locations, Pakistan
- Many Locations, Qatar
- Many Locations, Russia
- Many Locations, Saudi Arabia
- Many Locations, United Arab Emirates

REFERENCES:
- [Derived] Motaweih AK, Usova E, Hussain W, Dello Z, Schmidt B, Petri T. Effectiveness of combination therapy with nifedipine GITS: a prospective, 12-week observational study (AdADOSE). BMC Cardiovasc Disord. 2015 May 9;15:35. doi: 10.1186/s12872-015-0037-x. PMID 25956918